CLINICAL TRIAL: NCT00980954
Title: Phase III Randomized Study of Concurrent Chemotherapy and Pelvic Radiation Therapy With or Without Adjuvant Chemotherapy in High-Risk Patients With Early-Stage Cervical Carcinoma Following Radical Hysterectomy
Brief Title: Chemotherapy and Pelvic Radiation Therapy With or Without Additional Chemotherapy in Treating Patients With High-Risk Early-Stage Cervical Cancer After Radical Hysterectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0724; CDR0000654709; NCI-2011-01973 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RTOG 0724/GOG-0724 (Other: NRG Oncology)
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Results first posted 2024-11-06 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancer
Keywords: cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical squamous cell carcinoma; stage IA cervical cancer; stage IB cervical cancer; stage IIA cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Carboplatin; Cisplatin; Paclitaxel; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Cisplatin/Radiation Therapy (Active Comparator): Standard external beam radiation therapy (EBRT) or intensity-modulated radiation therapy (IMRT) to the pelvis once daily 5 days a week for 5-6 weeks as 45 Gy in 25 fractions or 50.4 Gy in 28 fractions (1.8 Gy/fraction). Concurrent cisplatin IV over one hour once weekly for 6 weeks as 40 mg/m^2, maximum dose 70 mg. A brachytherapy boost following radiation therapy is optional.
  Interventions: Drug: cisplatin; Radiation: intensity-modulated radiation therapy; Radiation: standard external beam radiation therapy; Radiation: Optional brachytherapy boost
- Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel (Experimental): Chemoradiotherapy as in arm I, followed 4-6 weeks later by paclitaxel IV [135 mg/m2, with maximum body surface area (BSA) of 2.0 m^2 over 3 hours] and carboplatin IV [area under the curve (AUC) 5 over 30 minutes] on day 1 of 21-day cycle for 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: cisplatin; Drug: paclitaxel; Radiation: intensity-modulated radiation therapy; Radiation: standard external beam radiation therapy; Radiation: Optional brachytherapy boost

INTERVENTIONS:
Drug: carboplatin — Intravenously
  Arms: Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel
Drug: cisplatin — Intravenously
Drug: paclitaxel — Intravenously
  Arms: Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel
Radiation: intensity-modulated radiation therapy — Daily fractions
  Other Names: IMRT
Radiation: standard external beam radiation therapy — Daily fractions
  Other Names: EBRT
Radiation: Optional brachytherapy boost — Low-dose rate (20-25 Gy single application) or high-dose rate (12-18 Gy 2-3 applications), dependent on external beam dose.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, paclitaxel, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. It is not yet known whether chemotherapy and radiation therapy are more effective when given with or without additional chemotherapy in treating cervical cancer.

PURPOSE: This randomized phase III trial is studying chemotherapy and pelvic radiation therapy to see how well they work when given with or without additional chemotherapy in treating patients with high-risk early-stage cervical cancer after radical hysterectomy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if administering adjuvant systemic chemotherapy after chemoradiotherapy will improve disease-free survival compared to chemoradiotherapy alone in patients with high-risk early-stage cervical carcinoma found to have positive nodes and/or positive parametria after radical hysterectomy.

Secondary

* To evaluate adverse events.
* To evaluate overall survival.
* To evaluate quality of life.
* To evaluate chemotherapy-induced neuropathy.
* To perform a post-hoc dose-volume evaluation between patients treated with standard radiotherapy and patients treated with intensity-modulated radiotherapy (IMRT) with respect to toxicity and local control.
* To collect fixed tissue samples to identify tumor molecular signatures that may be associated with patient outcomes, such as adverse events, disease-free survival, and overall survival.
* To collect blood samples to identify secreted factors from serum and plasma that may be associated with adverse events or outcome and to identify single nucleotide polymorphisms (SNPs) in genes from buffy coat that may be associated with a genetic predisposition to tumor formation itself or a response to cytotoxic therapy.

OUTLINE: This is a multicenter study. Patients are stratified according to planned use of brachytherapy (no vs. yes), radiotherapy modality - [standard external beam radiotherapy (EBRT) vs. intensity-modulated radiotherapy (IMRT)], and radiotherapy dose (45 Gy vs. 50.4 Gy). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo standard EBRT or IMRT to the pelvis once daily 5 days a week for 5-6 weeks. Patients also receive concurrent cisplatin IV over 1 hour once weekly for 6 weeks.

NOTE: Some patients may also undergo brachytherapy beginning within 7 days after completion of radiotherapy.

* Arm II: Patients receive chemoradiotherapy as in arm I. Beginning 4-6 weeks after completion of chemoradiotherapy, patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed by the Functional Assessment of Cancer Therapy - Gynecologic Oncology Group (FACT-GOG/NTX4), FACT-Cx, and FACIT-D questionnaires at baseline; at the completion of chemoradiotherapy; and then at 6, 12, and 24 months after completion of chemoradiotherapy.

Blood and tissue samples may be collected for gene expression analysis by immuno-histochemistry (IHC) and for biomarker and polymorphism studies.

After completion of study treatment, patients are followed up very 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous, adenosquamous, or adenocarcinoma of the cervix with any/all of the following high-risk features after surgery:

  * Positive pelvic nodes
  * Positive parametrium
  * Positive para-aortic nodes that have been completely resected and are positron emission tomography (PET)/computed tomography (CT) scan-negative

    * PET only required if positive para-aortic nodes during surgery
* Clinical stage IA2, IB, or IIA disease (this corresponds to surgical tumor node metastasis (TNM) staging of T1-T2, N1, M0)
* Must have undergone radical hysterectomy (open, laparoscopically, or robotic) and staging within the past 70 days

  * Para-aortic and pelvic node sampling required

    * If the patient did not have a para-aortic lymph node sampling/dissection, but had common iliac node dissection that was negative, a PET-CT is recommended, but not required
    * A negative pre- or post-operative PET scan or PET-CT scan of the para-aortic nodes is required if the patient did not undergo para-aortic or common iliac nodal sampling/dissection
  * No gross residual disease
* No neuroendocrine histology
* No distant metastases

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Absolute neutrophil count (ANC) ≥ 1,800/mm³
* Platelets ≥ 100,000/mm³
* White blood cell count (WBC) ≥ 4,000/mm³
* Hemoglobin ≥ 10.0 g/dL (transfusion or other intervention allowed)
* Serum creatinine ≤ 1.5 mg/dL
* Bilirubin ≤ 1.5 times upper limit of normal
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) normal
* Alkaline phosphatase normal
* Known HIV positivity allowed provided cluster of differentiation 4 (CD4) count is ≥ 350/mm³ within the past 14 days
* No other invasive malignancy within the past 3 years, except nonmelanomatous skin cancer or carcinoma in situ of the breast, oral cavity, or cervix
* No severe, active co-morbidity, including any of the following:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
  * Transmural myocardial infarction within the past 6 months
  * Acute bacterial or fungal infection requiring IV antibiotics at the time of study entry
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of study entry
  * Coagulation defects
* No prior allergic reaction to carboplatin, paclitaxel, and/or cisplatin

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior systemic chemotherapy for the current cervical cancer

  * Prior chemotherapy for a different cancer is allowed
* No prior radiotherapy to the pelvis that would result in overlap of radiotherapy fields

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2009-09; Primary Completion 2023-12-14 (Actual); Study Completion 2025-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anuja Jhingran, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (125):
- United States (119):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Providence Hospital, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mercy San Juan Medical Center, Carmichael, California
  - City of Hope Medical Center, Duarte, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Mercy Cancer Center, Sacramento, California
  - Mercy General Hospital Radiation Oncology Center, Sacramento, California
  - University of California At San Diego, San Diego, California
  - Saint Helena Hospital, St. Helena, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - University of Miami Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Memorial Healthcare System - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Jackson Memorial Hospital-Holtz Children's Hospital, Miami, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Grady Health System, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Joseph's-Candler Health System, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Saint Vincent Anderson Regional Hospital/Cancer Center, Anderson, Indiana
  - Saint Francis Hospital and Health Centers, Beech Grove, Indiana
  - Franciscan Saint Margaret Health-Hammond Campus, Hammond, Indiana
  - Franciscan Saint Francis Health-Indianapolis, Indianapolis, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kansas City Cancer Centers-Southwest, Overland Park, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Hickman Cancer Center, Adrian, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Kansas City Cancer Center - South, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Kansas City Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - The Nebraska Medical Center, Omaha, Nebraska
  - Elliot Hospital, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - UMDNJ - New Jersey Medical School, Newark, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Weiler Division, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Summa Health Center at Lake Medina, Medina, Ohio
  - UHHS-Chagrin Highlands Medical Center, Orange, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Robinson Radiation Oncology, Ravenna, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - Ireland Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Flower Hospital, Sylvania, Ohio
  - University of Toledo, Toledo, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Wheeling Hospital, Wheeling, West Virginia
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- McGill University Department of Oncology, Montreal, Quebec, Canada
- Pamela Youde Nethersole Eastern Hospital, Chai Wan, Hong Kong
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam, Kyeonggi-do
  - Seoul National University Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea Cancer Center Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I: Cisplatin/Radiation Therapy | Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel
Started | 118 | 118
Eligible | 109 | 103
Completed (Participants contributing data to results are considered to have completed the study.) | 109 | 103
Not Completed | 9 | 15
Not completed — Protocol Violation | 9 | 15

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Cisplatin/Radiation Therapy | Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel | Total
Number analyzed (Participants) | 109 | 103 | 212
Age, Customized [Median (Inter-Quartile Range); unit: years] | 47 [39 to 56] | 45 [38 to 56] | 46 [39 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 103 | 212
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 10 | 23
  Not Hispanic or Latino | 95 | 92 | 187
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 42 | 40 | 82
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 9 | 13
  White | 60 | 49 | 109
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 4 | 5
Zubrod performance status [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound; 5 = Death.
  Participants
    0 | 87 | 79 | 166
    1 | 22 | 24 | 46
Hysterectomy Procedure [Count of Participants; unit: Participants]
  Open | 64 | 54 | 118
  Laparoscopic | 26 | 22 | 48
  Robotic | 19 | 27 | 46
Histologic Type [Count of Participants; unit: Participants] — A description of a tumor based on how the cancer cells and tissue look under a microscope.
  Participants
    Squamous cell carcinoma | 88 | 74 | 162
    Adenosquamous carcinoma | 6 | 5 | 11
    Adenocarcinoma, not otherwise specificed (NOS) | 15 | 24 | 39
Histologic grade [Count of Participants; unit: Participants] — Histologic grade, also known as tumor grade, is a description of a tumor that's based on how abnormal the cancer cells and tissue look under a microscope, and how quickly the cancer cells are likely to grow and spread. It's used to help plan treatment and determine prognosis.
  Participants
    Gx-Grade cannot be assessed | 14 | 15 | 29
    G1-Well differentiated | 10 | 5 | 15
    G2-Moderately differentiated | 58 | 52 | 110
    G3-Poorly differentiated | 27 | 31 | 58
FIGO Staging (clinical) [AJCC 6th Edition] [Count of Participants; unit: Participants] — International Federation of Gynecology and Obstetrics (FIGO) staging is a system developed to stage (or measure) cancers that affect the female reproductive system, such as cervical, ovarian, and endometrial cancers. FIGO staging is based on three main factors: the size and extent of the tumor; the involvement of nearby lymph nodes; the presence or absence of distant metastases. The stages are numbered from I to IV, with subcategories represented by letters or numbers, indicating the severity and progression of the cancer, with lower numbers and letters indicating better prognosis.
  Participants
    IA2 | 3 | 6 | 9
    IB | 97 | 88 | 185
    IIA | 9 | 9 | 18
Pathologic T-Stage [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 6th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail with additional letters and numbers.
  Participants
    T0 | 2 | 1 | 3
    T1 | 1 | 2 | 3
    T1a1 | 1 | 1 | 2
    T1a2 | 2 | 6 | 8
    T1b | 4 | 8 | 12
    T1b1 | 39 | 34 | 73
    T1b2 | 23 | 15 | 38
    T2 | 6 | 10 | 16
    T2b | 30 | 24 | 54
    T3b | 1 | 2 | 3
Pathologic N-Stage [Count of Participants; unit: Participants] — Regional lymph nodes staging per American Joint Committee on Cancer (AJCC) 6th ed. refers to the number and/or extent of spread of lymph nodes that contain cancer. N0 means lymph nodes aren't involved. A higher number means the cancer is in more lymph nodes, farther away from the original tumor. NX means the lymph nodes cannot be assessed.
  Participants
    N0 | 30 | 26 | 56
    N1 | 79 | 77 | 156
Pathologic M-Stage [Count of Participants; unit: Participants] — Metastasis stage per the American Joint Committee on Cancer (AJCC) 6th ed. refers to the spread of the cancer to organs and tissues in other parts of the body. M0 = No distant metastasis; M1 = Distant metastasis; MX = Distant metastasis cannot be assessed.
  Participants
    M0 | 108 | 103 | 211
    M1 | 1 | 0 | 1
Positive Parametrium [Count of Participants; unit: Participants] — Cancer present.
  Participants
    No | 53 | 58 | 111
    Yes | 56 | 45 | 101
Positive Pelvic Nodes [Count of Participants; unit: Participants] — Cancer present.
  Participants
    No | 33 | 23 | 56
    Yes | 76 | 80 | 156
Positive Para-Aortic Nodes [Count of Participants; unit: Participants] — Cancer present.
  Participants
    No | 54 | 43 | 97
    Yes | 3 | 5 | 8
    Not sampled / dissected | 52 | 55 | 107
Intention to use brachytherapy [Count of Participants; unit: Participants]
  No | 61 | 58 | 119
  Yes | 48 | 45 | 93
Intended RT Modality [Count of Participants; unit: Participants]
  Standard RT | 46 | 41 | 87
  IMRT | 63 | 62 | 125
Intended RT Dose [Count of Participants; unit: Participants]
  45 Gy | 35 | 30 | 65
  50.4 Gy | 74 | 73 | 147

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (Percentage of Participants Alive Without Disease)
Description: Disease-free survival (DFS) is estimated by the Kaplan-Meier method. The distribution of DFS estimates between the two arms is compared using the log rank test. DFS time is measured from the date of randomization to the date of first DFS failure (local, regional or distant metastases failure or death due to any cause) or last follow-up (censored). Analysis was to occur after disease or death was reported for 50 participants.
Time Frame: From randomization to first failure (local, regional, or distant metastases failure or death due to any cause) or last follow-up. Maximum follow-up at the time of analysis was 12.8 years. The 2- and 4-year DFS estimates are reported.
Population: Eligible participants
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I: Cisplatin/Radiation Therapy | Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel
Number analyzed (Participants) | 109 | 103
percentage of participants
  2 years | 86.4 [80.8 to 92.0] | 82.1 [75.6 to 88.6]
  4 years | 76.2 [69.1 to 83.4] | 76.9 [69.6 to 84.3]
Statistical Analysis 1: Comparison: Arm I: Cisplatin/Radiation Therapy vs Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel; Sample size calculations are based on the primary hypothesis that 4 additional cycles of carboplatin and paclitaxel following concurrent radiation and weekly cisplatin will increase 4-year DFS from 80% to 90% for patients with cervical carcinoma with positive nodes and/or positive margins after a radical hysterectomy. One-sided alpha=0.05, statistical power=80%, 5.5 years of accrual with 4 years of follow-up, 2 interim significance tests. 50 DFS events are required to trigger this analysis; Test type: Superiority; p = 0.56, Log Rank — One-sided significance level = 0.05; Hazard Ratio (HR) = 1.05, 90% CI 2-sided [0.65 to 1.68] — Reference level = Arm I

2. Secondary Outcome: Overall Survival (Percentage of Participants Alive)
Description: Overall survival is estimated by the Kaplan-Meier method. The distribution of survival estimates between the two arms is compared using the log rank test. Survival time is measured from the date of randomization to the date of death from any cause or last known follow-up (censored). Analysis was to occur after disease or death was reported for 50 participants.
Time Frame: From randomization to death or last follow-up. Maximum follow-up time at time of analysis was 12.8 years. The 2- and 4-year survival estimates are reported.
Population: Eligible participants
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I: Cisplatin/Radiation Therapy | Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel
Number analyzed (Participants) | 109 | 103
percentage of participants
  2 years | 91.9 [87.4 to 96.4] | 91.4 [86.6 to 96.2]
  4 years | 87.3 [81.6 to 93.0] | 89.0 [83.5 to 94.4]
Statistical Analysis 1: Comparison: Arm I: Cisplatin/Radiation Therapy vs Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel; The 4-year overall survival rate for the control arm is expected to be approximately 85%. The overall survival will be compared between the two arms. The final targeted sample size of 235 patients with the longer accrual time, will provide 64% and 78% power to detect an increase in overall survival to 92% and 93% respectively, with a 1- sided alpha of 0.05; Test type: Superiority; p = 0.40, Log Rank — One-sided significance level = 0.05; Hazard Ratio (HR) = 0.91, 90% CI 2-sided [0.49 to 1.69]

3. Secondary Outcome: Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity (FACT/GOG-NTX) at 12 Months
Description: The FACT-GOG/NTX4 measures patient-reported symptoms of chemotherapy-induced peripheral neuropathy in cancer patients. Possible scores range from 0 to 16 with higher scores indicating a better condition. Analysis of covariance, using the baseline score as a covariate, will be used to determine if there is a difference between the treatment arms.
Time Frame: Baseline and 12 months after the completion of concurrent chemoradiation (6 weeks)
Reporting Status: Not Posted, anticipated posting 2026-09

4. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Diarrhea (FACIT-D) Diarrhea Subscore at 12 Months
Description: The diarrhea-specific subscore of the FACIT-D measures patient-reported diarrhea symptoms. Possible scores range from 0 to 44 with higher scores indicating a better quality of life. Analysis of covariance, using the baseline score as a covariate, will be used to determine if there is a difference between the treatment arms.
Time Frame: Baseline and 12 months after the completion of concurrent chemoradiation (6 weeks)
Reporting Status: Not Posted, anticipated posting 2026-09

5. Secondary Outcome: Functional Assessment of Cancer Therapy - Cervix (FACT-Cx) Cervical Cancer Subscore at 12 Months
Description: The cervical cancer subscore of the FACT-Cx measures patient-reported symptoms and problems related to cervical cancer. Possible scores range from 0 to 60 with higher scores indicating a better quality of life. Analysis of covariance, using the baseline score as a covariate, will be used to determine if there is a difference between the treatment arms.
Time Frame: Baseline and 12 months after the completion of concurrent chemoradiation (6 weeks)
Reporting Status: Not Posted, anticipated posting 2026-09

6. Secondary Outcome: Number of Participants by Highest Grade Adverse Event Reported
Description: Common Terminology Criteria for Adverse Events (version 4.0) grades adverse event severity as follows: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = death related to adverse event. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: From randomization to the date of last known follow-up. Maximum follow-up time was 12.8 years.
Population: Eligible participants who started protocol treatment and were assessed for adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Cisplatin/Radiation Therapy | Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel
Number analyzed (Participants) | 107 | 101
Participants
  Grade 1 | 13 | 4
  Grade 2 | 43 | 30
  Grade 3 | 39 | 44
  Grade 4 | 8 | 21
  Grade 5 | 0 | 0

7. Secondary Outcome: Associations Between Tumor Molecular Signatures, From Fixed Tissue, and Outcomes Such as Adverse Events, Disease Free Survival and Overall Survival
Time Frame: From randomization to last follow-up
Population: The protocol did not provide sufficient detail to meet current National Cancer Institute requirements for release of specimens from the NRG Oncology tissue bank for the protocol-specified objective, therefore no assays were performed, and no data were collected for this outcome measure. Specimen use will require federal approval and funding separate from this trial.
Arm/Group | Arm I: Cisplatin/Radiation Therapy | Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Associations Between Secreted Factors From Serum and Plasma With Adverse Events or Outcome
Time Frame: From randomization to last follow-up.
Population: as for outcome 7
Arm/Group | Arm I: Cisplatin/Radiation Therapy | Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Associations Between Single Nucleotide Polymorphisms (SNPs) in Genes From Buffy Coat and a Genetic Predisposition to Tumor Formation Itself or a Response to Cytotoxic Therapy
Time Frame: From randomization to last follow-up.
Population: as for outcome 7
Arm/Group | Arm I: Cisplatin/Radiation Therapy | Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Disease-free Survival (Percentage of Participants Alive Without Disease) by Ethnicity
Description: NIH-required analysis. Disease-free survival (DFS) is estimated by the Kaplan-Meier method. The distribution of DFS estimates between the two arms is compared using the log rank test. DFS time is measured from the date of randomization to the date of first DFS failure (local, regional or distant metastases failure or death due to any cause) or last follow-up (censored). Analysis was to occur after disease or death was reported for 50 participants.
Time Frame: as for outcome 1
Population: Eligible participants stratified by ethnicity
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I: Cisplatin/Radiation Therapy | Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel
Number analyzed (Participants) | 109 | 103
percentage of participants
  Hispanic or Latino: 2 years: number analyzed (Participants) | 13 | 10
  Hispanic or Latino: 2 years | 83.9 [66.7 to 100.0] | 77.8 [55.0 to 100.0]
  Hispanic or Latino: 4 years: number analyzed (Participants) | 13 | 10
  Hispanic or Latino: 4 years | 83.9 [66.7 to 100.0] | 64.8 [37.6 to 92.0]
  Not Hispanic or Latino: 2 years: number analyzed (Participants) | 95 | 92
  Not Hispanic or Latino: 2 years | 86.7 [80.9 to 92.6] | 83.4 [76.7 to 90.1]
  Not Hispanic or Latino: 4 years: number analyzed (Participants) | 95 | 92
  Not Hispanic or Latino: 4 years | 75.4 [67.7 to 83.1] | 79.0 [71.5 to 86.5]
  Unknown or Not Reported: 2 years: number analyzed (Participants) | 1 | 1
  Unknown or Not Reported: 2 years | NA [NA to NA] — Cannot be calculated because the participant was censored prior to the timepoint. | 0 [0 to 100]
  Unknown or Not Reported: 4 years: number analyzed (Participants) | 1 | 1
  Unknown or Not Reported: 4 years | NA [NA to NA] — Cannot be calculated because the participant was censored prior to the timepoint. | 0 [0 to 100]

11. Other Pre Specified Outcome: Disease-free Survival (Percentage of Participants Alive Without Disease) by Race
Description: as for outcome 10
Time Frame: as for outcome 1
Population: Eligible participants stratified by race
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I: Cisplatin/Radiation Therapy | Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel
Number analyzed (Participants) | 109 | 103
percentage of participants
  American Indian or Alaska Native: 2 years: number analyzed (Participants) | 1 | 1
  American Indian or Alaska Native: 2 years | 100 [NA to NA] — SAS software does not compute a confidence interval when the estimate is 100%. | 100 [NA to NA] — SAS software does not compute a confidence interval when the estimate is 100%.
  American Indian or Alaska Native: 4 years: number analyzed (Participants) | 1 | 1
  American Indian or Alaska Native: 4 years | NA [NA to NA] — Cannot be calculated because the participant was censored prior to the timepoint. | NA [NA to NA] — Cannot be calculated because the participant was censored prior to the timepoint.
  Asian: 2 years: number analyzed (Participants) | 42 | 40
  Asian: 2 years | 87.1 [78.2 to 96.0] | 74.4 [62.3 to 86.6]
  Asian: 4 years: number analyzed (Participants) | 42 | 40
  Asian: 4 years | 76.0 [64.5 to 87.5] | 64.2 [50.3 to 78.0]
  Black or African American: 2 years: number analyzed (Participants) | 4 | 9
  Black or African American: 2 years | 100 [NA to NA] — SAS software does not compute a confidence interval when the estimate is 100%. | 87.5 [68.3 to 100.0]
  Black or African American: 4 years: number analyzed (Participants) | 4 | 9
  Black or African American: 4 years | 100 [NA to NA] — SAS software does not compute a confidence interval when the estimate is 100%. | 87.5 [68.3 to 100.0]
  White: 2 years: number analyzed (Participants) | 60 | 49
  White: 2 years | 85.9 [78.3 to 93.5] | 89.3 [81.8 to 96.7]
  White: 4 years: number analyzed (Participants) | 60 | 49
  White: 4 years | 75.4 [65.5 to 85.3] | 86.6 [78.1 to 95.0]
  More than one race: 2 years: number analyzed (Participants) | 1 | 0
  More than one race: 2 years | 100 [NA to NA] — SAS software does not compute a confidence interval when the estimate is 100% |
  More than one race: 4 years: number analyzed (Participants) | 1 | 0
  More than one race: 4 years | NA [NA to NA] — Cannot be calculated because the participant was censored prior to the timepoint. |
  Unknown or Not Reported: 2 years: number analyzed (Participants) | 1 | 4
  Unknown or Not Reported: 2 years | 0 [0 to 100] | 50 [8.9 to 91.1]
  Unknown or Not Reported: 4 years: number analyzed (Participants) | 1 | 4
  Unknown or Not Reported: 4 years | 0 [0 to 100] | 50 [8.9 to 91.1]

ADVERSE EVENTS:
Time Frame: From randomization to the date of last known follow-up. Maximum follow-up time was 12.8 years.
Description: All-cause mortality was assessed in eligible participants. Adverse events were assessed in eligible participants who started protocol treatment were assessed for adverse events.
Arm/Group | Arm I: Cisplatin/Radiation Therapy | Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel
All-Cause Mortality (participants affected / at risk) | 17/109 | 13/103
Serious Adverse Events (participants affected / at risk) | 14/107 | 25/101
Other Adverse Events (participants affected / at risk) | 103/107 | 99/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Cisplatin/Radiation Therapy (N=107) | Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel (N=101)
Anemia (Blood and lymphatic system disorders) | 3 | 3
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 3
Diarrhea (Gastrointestinal disorders) | 2 | 5
Gastritis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2
Fever (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 1 | 2
Tooth infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 4
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 1
Creatinine increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 2
Neutrophil count decreased (Investigations) | 1 | 2
Platelet count decreased (Investigations) | 1 | 2
White blood cell decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Cisplatin/Radiation Therapy (N=107) | Arm II: Cisplatin/Radiation Therapy + Carboplatin/Paclitaxel (N=101)
Anemia (Blood and lymphatic system disorders) | 48 | 60
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 10 | 7
Chest pain - cardiac (Cardiac disorders) | 3 | 6
Hearing impaired (Ear and labyrinth disorders) | 3 | 6
Tinnitus (Ear and labyrinth disorders) | 19 | 21
Blurred vision (Eye disorders) | 5 | 8
Abdominal pain (Gastrointestinal disorders) | 32 | 31
Anal pain (Gastrointestinal disorders) | 4 | 9
Constipation (Gastrointestinal disorders) | 40 | 54
Diarrhea (Gastrointestinal disorders) | 62 | 57
Dyspepsia (Gastrointestinal disorders) | 16 | 19
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 | 5
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 8 | 7
Mucositis oral (Gastrointestinal disorders) | 3 | 7
Nausea (Gastrointestinal disorders) | 71 | 70
Vomiting (Gastrointestinal disorders) | 27 | 34
Chills (General disorders) | 6 | 3
Edema limbs (General disorders) | 12 | 5
Fatigue (General disorders) | 58 | 59
Fever (General disorders) | 7 | 11
General disorders and administration site conditions - Other, specify (General disorders) | 4 | 7
Pain (General disorders) | 21 | 16
Infections and infestations - Other, specify (Infections and infestations) | 4 | 6
Urinary tract infection (Infections and infestations) | 10 | 20
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 6
Alanine aminotransferase increased (Investigations) | 11 | 18
Aspartate aminotransferase increased (Investigations) | 5 | 8
Creatinine increased (Investigations) | 8 | 12
Lymphocyte count decreased (Investigations) | 17 | 22
Neutrophil count decreased (Investigations) | 35 | 52
Platelet count decreased (Investigations) | 28 | 34
Weight gain (Investigations) | 2 | 7
Weight loss (Investigations) | 8 | 10
White blood cell decreased (Investigations) | 45 | 52
Anorexia (Metabolism and nutrition disorders) | 27 | 36
Hyperglycemia (Metabolism and nutrition disorders) | 10 | 17
Hypernatremia (Metabolism and nutrition disorders) | 0 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 11
Hypokalemia (Metabolism and nutrition disorders) | 12 | 12
Hypomagnesemia (Metabolism and nutrition disorders) | 19 | 22
Hyponatremia (Metabolism and nutrition disorders) | 12 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 12
Dizziness (Nervous system disorders) | 12 | 11
Dysgeusia (Nervous system disorders) | 3 | 10
Headache (Nervous system disorders) | 18 | 29
Paresthesia (Nervous system disorders) | 5 | 19
Peripheral motor neuropathy (Nervous system disorders) | 3 | 10
Peripheral sensory neuropathy (Nervous system disorders) | 22 | 49
Anxiety (Psychiatric disorders) | 13 | 19
Depression (Psychiatric disorders) | 6 | 9
Insomnia (Psychiatric disorders) | 12 | 20
Cystitis noninfective (Renal and urinary disorders) | 2 | 12
Hematuria (Renal and urinary disorders) | 2 | 7
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 13 | 8
Urinary frequency (Renal and urinary disorders) | 17 | 23
Urinary incontinence (Renal and urinary disorders) | 7 | 11
Urinary retention (Renal and urinary disorders) | 7 | 11
Urinary tract pain (Renal and urinary disorders) | 8 | 22
Urinary urgency (Renal and urinary disorders) | 8 | 8
Dyspareunia (Reproductive system and breast disorders) | 10 | 12
Pelvic pain (Reproductive system and breast disorders) | 10 | 20
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 4 | 9
Vaginal discharge (Reproductive system and breast disorders) | 8 | 8
Vaginal dryness (Reproductive system and breast disorders) | 9 | 8
Vaginal hemorrhage (Reproductive system and breast disorders) | 3 | 9
Vaginal pain (Reproductive system and breast disorders) | 4 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 17
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 37
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 7
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 10 | 5
Hot flashes (Vascular disorders) | 22 | 22
Hypertension (Vascular disorders) | 9 | 7
Lymphedema (Vascular disorders) | 9 | 10
Thromboembolic event (Vascular disorders) | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT00980954/Prot_SAP_001.pdf
  • Informed Consent Form (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT00980954/ICF_000.pdf